CLINICAL TRIAL: NCT04559126
Title: A Randomized, Double-Blind, Placebo-Controlled, First-In-Human Study of Orally Administered EDP-297 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (SAD), Multiple Ascending Doses (MAD), and the Effect of Food on EDP-297 Pharmacokinetics in Healthy Subjects
Brief Title: A Study of EDP-297 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 297-001
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: NASH - Nonalcoholic Steatohepatitis With Liver Fibrosis
Keywords: "First-in-Human"; Single Ascending Dose; Multiple Ascending Dose; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- EDP-297 SAD Cohorts (Experimental): EDP-297 Dose 1, Dose 2, Dose 3, Dose 4, Dose 5 and Dose 6 oral solution, once daily in one single administration
  Interventions: Drug: EDP-297
- EDP-297 MAD Cohorts (Experimental): EDP-297 Dose 1, Dose 2 and Dose 3 oral solution, once daily for 14 days
  Interventions: Drug: EDP-297
- EDP-297 SAD Placebo Cohort (Placebo Comparator): Matching placebo, oral solution, once daily in one single administration
  Interventions: Drug: Placebo
- EDP-297 MAD Placebo Cohort (Placebo Comparator): Matching placebo, oral solution, once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-297 — EDP-297 Oral solution
  Arms: EDP-297 MAD Cohorts; EDP-297 SAD Cohorts
Drug: Placebo — placebo to match EDP-297
  Arms: EDP-297 MAD Placebo Cohort; EDP-297 SAD Placebo Cohort

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study. It will assess the safety, tolerability, and pharmacokinetics of orally administered single and multiple doses of EDP-297 in healthy adult subjects.

DETAILED DESCRIPTION:
The first phase assesses single ascending doses of EDP-297 or placebo in healthy subjects. A "fasted" and "fed" two-part cohort will also assess food effect.

The second phase assesses multiple ascending doses of EDP-297 or placebo for 14-days in healthy subjects.

Each cohort within each phase will enroll a total of 8 subjects who will be randomized to receive EDP-297 or placebo. The cohort assessing food effect will enroll 10 subjects randomized to receive EDP-297 or placebo

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -2.
* Current tobacco smokers or use of tobacco within 1 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption exceeding 14 drinks/week for females and 21 drinks/week for males within 6 months of Screening.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 8 Days in SAD Cohorts
Safety measured by adverse events | Up to 21 Days in MAD Cohorts

SECONDARY OUTCOMES:
Cmax of EDP-297 | Up to 6 Days in SAD Cohorts
Cmax of EDP-297 | Up to 18 Days in MAD Cohorts
AUC of EDP-297 | Up to 6 Days in SAD Cohorts
AUC of EDP-297 | Up to 18 Days in MAD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

REFERENCES:
- [Derived] Marotta C, Ahmad A, Luo E, Oosterhaven J, van Marle S, Adda N. EDP-297: A novel, farnesoid X receptor agonist-Results of a phase I study in healthy subjects. Clin Transl Sci. 2023 Feb;16(2):338-351. doi: 10.1111/cts.13453. Epub 2022 Nov 21. PMID 36369848